CLINICAL TRIAL: NCT00546858
Title: Part A: STUDY OF THE RELATIONSHIP OF INTERSTITIAL CYSTITIS TO VULVODYNIA
Brief Title: Relationship of Interstitial Cystitis to Vulvodynia
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Other Study IDs: 2007-183
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Interstitial Cystitis
Keywords: Pelvic pain; Vulvar pain
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain; Vulvodynia | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey: Patients with interstitial cystitis
  Interventions: Other: Physical Examination

INTERVENTIONS:
Other: Physical Examination — Patients will be invited to be evaluated in the Urology Research office at a future date.

SUMMARY:
This study is important in urologic nursing since many patients have interstitial cystitis (IC), a condition of frequency, urgency and pain affecting more than 1 million women in the United States. The vulva may actually be the site of some of the reported pain in women with IC, not the urethra or bladder. IC and vulvodynia can impact one's sexual functioning and diminish one's quality of life.

The purpose of this two-part study is to identify and clinically confirm the presence of vulvodynia in women diagnosed with Interstitial Cystitis (IC).

ELIGIBILITY:
Inclusion Criteria:

* Females who are 18 years of age and older.
* Diagnosis of interstitial cystitis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of Interstitial Cystitis from the practices of Dr Ananias Diokno and Dr Kenneth Peters will be mailed a survey.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The purpose of this two-part study is to identify and clinically confirm the presence of vulvodynia in women diagnosed with Interstitial Cystitis (IC). | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: Donna Carrico, NP, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States